CLINICAL TRIAL: NCT05418751
Title: Effectiveness of a Manual Therapy Protocol on Women With Pelvic Pain Due to Endometriosis: a Randomised Clinical Trial
Brief Title: Effectiveness of a Manual Therapy Protocol on Women With Pelvic Pain Due to Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Marta Inglés de la Torre, Professor, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 19866206
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Endometriosis; Pelvic Pain
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy group (Experimental): Patients in this group (n=20) will receive a manual therapy protocol.
  Interventions: Other: Manual therapy
- Placebo group (Placebo Comparator): Patients in this group (n=20) will receive a placebo treatment.
  Interventions: Other: Placebo treatment

INTERVENTIONS:
Other: Manual therapy — Participants will received a manual therapy protocol consisting of the following techniques: manipulation of the occipito-atlanto-axial joint (C0-C1-C2), suboccipital inhibition technique, manipulation of the thoracolumbar hinge (T12-L1), global manipulation of the bilateral pelvis, global abdominal hemodynamic technique, functional technique of the pelvic diaphragm and stretching of the lumbopelvic musculature.
  Arms: Manual therapy group
Other: Placebo treatment — Participants will receive light contact on the same points and for the same amount of time as the experimental group, with no intention to treat.
  Arms: Placebo group

SUMMARY:
Endometriosis is a debilitating disease with features of chronic inflammation that affects 10-15% of women of reproductive age. Pelvic pain is one of the most common symptoms in women with endometriosis, and many of them report that it affects their quality of life. In addition, women with endometriosis, especially those with pelvic pain, also have an increased vulnerability to various psychiatric disorders, such as depression and anxiety.

In this context, physical therapy can contribute to the multidisciplinary assessment and treatment of pelvic pain. In addition, manual therapy could improve certain variables related to central sensitization, such as inhibitory pain regulation and neuronal excitability in the dorsal horn of the medulla, in patients with chronic pain. Some prospective studies have applied manual therapy in patients with pelvic pain due to endometriosis, and have shown a trend towards improvement of pain and quality of life. Moreover, it is considered a well-tolerated and accepted treatment by patients.

However, to date, it has not been investigated whether the application of a manual therapy protocol improves pelvic pain and other endometriosis-associated symptoms, lumbar mobility, medication intake, depression and anxiety levels, and quality of life in women with endometriosis-associated pelvic pain compared to a placebo treatment.

DETAILED DESCRIPTION:
Endometriosis is a debilitating disease with features of chronic inflammation that affects 10-15% of women of reproductive age. Pelvic pain is one of the most common symptoms in women with endometriosis, and many of them report that it affects their quality of life. In addition, women with endometriosis, especially those with pelvic pain, also have an increased vulnerability to various psychiatric disorders, such as depression and anxiety.

In this context, physical therapy can contribute to the multidisciplinary assessment and treatment of pelvic pain. In addition, manual therapy could improve certain variables related to central sensitization, such as inhibitory pain regulation and neuronal excitability in the dorsal horn of the medulla, in patients with chronic pain. Some prospective studies have applied manual therapy in patients with pelvic pain due to endometriosis, and have shown a trend towards improvement of pain and quality of life. Moreover, it is considered a well-tolerated and accepted treatment by patients.

However, to date, it has not been investigated whether the application of a manual therapy protocol improves pelvic pain and other endometriosis-associated symptoms, lumbar mobility, medication intake, depression and anxiety levels, and quality of life in women with endometriosis-associated pelvic pain compared to a placebo treatment.

Therefore, this is a randomized clinical trial in which two groups of twenty people in each group will participate, with different interventions:

* Experimental group: manual therapy protocol.
* Placebo group: placebo treatment. Participants will be evaluated in four moments, at baseline, post-intervention, 1-month follow-up and 6-month follow-up.

Data analysis will be performed with SPSS statistic program (v24). Normality and homoscedasticity will be analyzed by Shapiro-Wilk t-test and Levene test, respectively. Multifactorial ANOVA will be performed with two groups (experimental and placebo group) and four-time assessments. For comparation between groups Bonferroni will be used. When p<0.05 statistically significant differences will be assumed.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal woman aged between 18 and 50 years.
* Diagnosis of endometriosis and associated pelvic pain.

Exclusion Criteria:

* Being pregnant.
* Having rheumatic or degenerative neurological diseases, as well as any other injury or disease that causes pelvic pain.
* Any pelvic surgery of less than one year of evolution (for example, cesarean sections).
* Having received physical therapy treatment within the last three months.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Endometriosis symptoms. The endometriosis health profile questionnaire (EHP-30Q) | 5 minutes
  5-point Likert scale, where 0=never, 1=rarely, 2=sometimes, 3=often, and 4=always. Raw scores for the questions within a scale are summed and transformed to a 0-100 scale, with higher scores indicating worse health-related quality of life.

SECONDARY OUTCOMES:
Health related quality of life. 36-Item Short Form Survey (SF-36) | 5 minutes
  From 0 to 100 points. Higher scores mean a better outcome.
Lumbar range of movement. Modified Schober Test | 5 minutes
  Higher scores mean a better outcome.< 2cm indicates severe restriction in lumbar flexion, 2-4 cm indicates moderate restriction and >4 cm indicates without restriction.
Depression. Beck Depression Index (BDI-II) | 5 minutes
  From 0 to 21 points. Higher scores mean greater depression.
Anxiety. State Trait Anxiety Index (STAI) | 5 minutes
  Scores range from 20 to 80, with higher scores correlating with greater anxiety.
Medication intake. Diary | 8 months
  Name of the drug, dosage and frequency of intake.
Impression of change after treatment. Patient global Perception of Change Scale (PGICS) | 1 minute
  From 1 to 7. Scale where 7=very much improved, 6= much improved, 5=minimally improved, 4=no change, 3=minimally worse, 2=much worse, 1=very much worse."

CONTACTS AND LOCATIONS:
Overall Officials: Marta Inglés, PhD, Principal Investigator — University of Valencia
Locations (1):
- Faculty of Physiotherapy, University of Valencia, Valencia, Spain

REFERENCES:
- [Background] Aredo JV, Heyrana KJ, Karp BI, Shah JP, Stratton P. Relating Chronic Pelvic Pain and Endometriosis to Signs of Sensitization and Myofascial Pain and Dysfunction. Semin Reprod Med. 2017 Jan;35(1):88-97. doi: 10.1055/s-0036-1597123. Epub 2017 Jan 3. PMID 28049214
- [Background] Arribas-Romano A, Fernandez-Carnero J, Molina-Rueda F, Angulo-Diaz-Parreno S, Navarro-Santana MJ. Efficacy of Physical Therapy on Nociceptive Pain Processing Alterations in Patients with Chronic Musculoskeletal Pain: A Systematic Review and Meta-analysis. Pain Med. 2020 Oct 1;21(10):2502-2517. doi: 10.1093/pm/pnz366. PMID 32100027
- [Background] Berghmans B. Physiotherapy for pelvic pain and female sexual dysfunction: an untapped resource. Int Urogynecol J. 2018 May;29(5):631-638. doi: 10.1007/s00192-017-3536-8. Epub 2018 Jan 9. PMID 29318334
- [Background] Sillem M, Juhasz-Boss I, Klausmeier I, Mechsner S, Siedentopf F, Solomayer E. Osteopathy for Endometriosis and Chronic Pelvic Pain - a Pilot Study. Geburtshilfe Frauenheilkd. 2016 Sep;76(9):960-963. doi: 10.1055/s-0042-111010. PMID 27681520
- [Background] Zullo F, Spagnolo E, Saccone G, Acunzo M, Xodo S, Ceccaroni M, Berghella V. Endometriosis and obstetrics complications: a systematic review and meta-analysis. Fertil Steril. 2017 Oct;108(4):667-672.e5. doi: 10.1016/j.fertnstert.2017.07.019. Epub 2017 Sep 2. PMID 28874260